CLINICAL TRIAL: NCT00311584
Title: A Phase II Study of Irinotecan + Temozolomide in Children With Recurrent Neuroblastoma
Brief Title: Irinotecan and Temozolomide in Treating Young Patients With Recurrent Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANBL0421; CDR0000465487 (Other: Clinical Trials.gov); COG-ANBL0421 (Other: Children's Oncology Group)
Record Dates: First submitted 2006-04-05; First posted 2006-04-06 (Estimated); Results first posted 2014-01-16 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-09

CONDITIONS: Neuroblastoma
Keywords: recurrent neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Irinotecan; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Disease measurable by CT or MRI scan (Irinotecan/Temozolomide) (Experimental): Measurable by CT scan (Computed Tomography) or MRI scan (Magnetic Resonance Imaging). Patients receive irinotecan hydrochloride IV (10 mg/m2/dose) over 1 hour on days 1-5 and 8-12 and oral temozolomide (100 mg/m2/dose) on days 1-5. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: irinotecan hydrochloride; Drug: temozolomide
- Disease eval by bone marrow or MIBG (Irinotecan/Temozolomide) (Experimental): Evaluation by bone marrow or MIBG scan (metaiodobenzylguanidine scan, a radiopharmaceutical). Patients receive irinotecan hydrochloride IV (10 mg/m2/dose) over 1 hour on days 1-5 and 8-12 and oral temozolomide (100 mg/m2/dose) on days 1-5. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: irinotecan hydrochloride; Drug: temozolomide

INTERVENTIONS:
Drug: irinotecan hydrochloride — Given IV
  Other Names: CPT-11; NSC #616348
Drug: temozolomide — Given IV
  Other Names: TEMODAR; NSC #362856

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan and temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving irinotecan together with temozolomide works in treating young patients with recurrent neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in pediatric patients with relapsed neuroblastoma (NB) treated with irinotecan hydrochloride and temozolomide.
* Determine the toxicities associated with irinotecan and temozolomide in patients treated with this regimen.

Secondary

* Evaluate the impact of p53 loss of function on response rate and event-free survival from start of relapse therapy.
* Collect data for ongoing analyses of UGT1A1 polymorphisms in these patients.
* Collect and bank serum and nucleic acid specimen to facilitate future biomarker studies.
* Evaluate the feasibility of collecting blood samples on a group wide basis for assessment of changes in circulating markers of angiogenesis.
* Assess, preliminarily, the effects of irinotecan hydrochloride and temozolomide on circulating markers of angiogenesis.

OUTLINE: This is a multicenter study.

Patients are stratified according to disease status (measurable disease [measured by conventional CT scan and/or MRI] vs evaluable disease [tumor detected by conventional morphologic analysis of bone marrow aspirate/biopsy AND/OR abnormal uptake at ≥ 1 site on MIBG scan]).

Patients receive irinotecan hydrochloride IV over 1 hour on days 1-5 and 8-12 and oral temozolomide on days 1-5. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 10 years.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed neuroblastoma AND/OR demonstration of tumor cells in the bone marrow with increased urinary catecholamines at initial diagnosis

  * Patients with elevated catecholamines only are not eligible
* Meets 1 of the following criteria:

  * Recurrent disease following aggressive, multidrug, frontline chemotherapy, defined as chemotherapy given with ≥ 2 agents, including an alkylating agent and a platinum-containing compound
  * Resistant/refractory disease during aggressive, multidrug, frontline chemotherapy
* Must meet 1 of the following criteria for documentation of disease:

  * Unidimensionally measurable tumor ≥ 20 mm by MRI (Magnetic Resonance Imaging), CT scan (Computed Tomography), or x-ray OR ≥ 10 mm by spiral CT scan within 4 weeks prior to study entry

    * Patients with residual stable tumor upon completion of frontline therapy must undergo biopsy to document presence of a viable neuroblastoma
    * If the measurable target lesion was previously radiated, a biopsy must be performed ≥ 4 weeks after radiation was completed AND the biopsy must demonstrate viable neuroblastoma
  * MIBG scan (metaiodobenzylguanidine scan, a radiopharmaceutical) with positive uptake at ≥ 1 site within 4 weeks prior to study entry

    * Patients with residual stable MIBG-positive lesions upon completion of frontline therapy must undergo biopsy to document presence of viable neuroblastoma
    * If the patient has only 1 MIBG-positive lesion, and that lesion was previously radiated, a biopsy must be performed ≥ 4 weeks after radiation was completed AND the biopsy must demonstrate viable neuroblastoma
  * Bone marrow with tumor cells on routine morphology (not by neuron-specific enolase staining only) of bilateral aspirate and/or biopsy on 1 bone marrow sample within 2 weeks prior to study entry
* No extensive marrow disease
* No myelodysplastic syndrome

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) 50-100% (for patients > 16 years of age) OR Lansky PS 50-100% (for patients ≤ 16 years of age)
* Life expectancy ≥ 8 weeks
* Absolute neutrophil count ≥ 750/mm^3
* Platelet count ≥ 75,000/mm^3 (transfusion independent)
* Hemoglobin ≥ 8.5 mg/dL (transfusion allowed)
* Creatinine adjusted according to age as follows:

  * No greater than 0.4 mg/dL (≤ 5 months)
  * No greater than 0.5 mg/dL (6 months -11 months)
  * No greater than 0.6 mg/dL (1 year-23 months)
  * No greater than 0.8 mg/dL (2 years-5 years)
  * No greater than 1.0 mg/dL (6 years-9 years)
  * No greater than 1.2 mg/dL (10 years-12 years)
  * No greater than 1.4 mg/dL (13 years and over [female])
  * No greater than 1.5 mg/dL (13 years to 15 years [male])
  * No greater than 1.7 mg/dL (16 years and over [male]) OR
* Creatinine clearance or radioisotope glomerular filtration rate at least 70 mL/min
* Bilirubin ≤ 1.5 times upper limit of normal (ULN) for age
* ALT < 2.5 times ULN for age
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Seizure disorder allowed provided seizures are well controlled on non-EIAC medication
* No active diarrhea or uncontrolled infection
* No other malignancy, including secondary malignancy

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior front-line therapy (e.g., surgery, chemotherapy, immunotherapy, radiotherapy, or retinoids) allowed
* Recovered from prior therapy
* More than 4 weeks since prior radiation therapy to the site of any lesion that will be identified as a target lesion to measure tumor response
* At least 2 weeks since prior myelosuppressive therapy (4 weeks for nitrosourea)
* At least 1 week since prior therapy with an antineoplastic biologic agent or retinoid
* At least 1 week since prior growth factors
* At least 1 week since prior and no other concurrent anticancer agents
* At least 1 week since prior and no concurrent enzyme-inducing anticonvulsants (EIAC), including phenytoin, phenobarbital, valproic acid, or carbamazepine

  * Concurrent gabapentin or levetiracetam allowed
* Concurrent palliative radiation therapy to sites not used to measure tumor response allowed
* No prior allogeneic stem cell transplantation (SCT)

  * Prior autologous SCT allowed
* No prior second-line chemotherapy for relapsed or refractory disease
* No concurrent immunomodulating agents

  * Concurrent steroids for transfusion/infusion reactions or for treatment of edema associated with CNS lesions allowed

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 2006-04; Primary Completion 2009-03 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rochelle Bagatell, MD, Study Chair — University of Arizona; Cynthia S. Kretschmar, MD, Study Chair — Floating Hospital for Children at Tufts - New England Medical Center
Locations (128):
- United States (110):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama - Birmingham, Birmingham, Alabama
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Sutter Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center - Oakland, Sacramento, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Stanford Cancer Center, Stanford, California
  - Children's Hospital Center for Cancer and Blood Disorders, Aurora, Colorado
  - Carole and Ray Neag Comprehensive Cancer Center at the University of Connecticut Health Center, Farmington, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - University of Illinois Cancer Center, Chicago, Illinois
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Floating Hospital for Children at Tufts - New England Medical Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Children's Hospital, Omaha, Nebraska
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Overlook Hospital, Morristown, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Maimonides Cancer Center at Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Medical Center - Dayton, Dayton, Ohio
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (5):
  - John Hunter Hospital, Newcastle, New South Wales
  - Westmead Institute for Cancer Research at Westmead Hospital, Westmead, New South Wales
  - Royal Children's Hospital, Brisbane, Queensland
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (13):
  - University of Alberta Hospital, Edmonton, Alberta
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan
  - Centre Hospitalier Universitaire de Quebec, Québec

REFERENCES:
- [Result] Bagatell R, London WB, Wagner LM, Voss SD, Stewart CF, Maris JM, Kretschmar C, Cohn SL. Phase II study of irinotecan and temozolomide in children with relapsed or refractory neuroblastoma: a Children's Oncology Group study. J Clin Oncol. 2011 Jan 10;29(2):208-13. doi: 10.1200/JCO.2010.31.7107. Epub 2010 Nov 29. PMID 21115869

RESULTS

PARTICIPANT FLOW:
Groups:
- Disease Eval by Bone Marrow or MIBG (Irinotecan/Temozolomide): Evaluation by bone marrow or MIBG scan (metaiodobenzylguanidine scan, a radiopharmaceutical). Patients receive irinotecan hydrochloride IV (10 mg/m2/dose) over 1 hour on days 1-5 and 8-12 and oral temozolomide (100 mg/m2/dose) on days 1-5. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  irinotecan hydrochloride : Given IV
  temozolomide : Given IV
- Disease Measurable by CT or MRI Scan (Irinotecan/Temozolomide): Measurable by CT scan (Computed Tomography) or MRI scan (Magnetic Resonance Imaging). Patients receive irinotecan hydrochloride (10 mg/m2/dose) over 1 hour on days 1-5 and 8-12 and oral temozolomide (100 mg/m2/dose) on days 1-5. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  irinotecan hydrochloride : Given IV
  temozolomide : Given IV
Period: Overall Study
Arm/Group | Disease Eval by Bone Marrow or MIBG (Irinotecan/Temozolomide) | Disease Measurable by CT or MRI Scan (Irinotecan/Temozolomide)
Started | 29 | 30
Completed | 9 | 7
Not Completed | 20 | 23
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 12 | 15
Not completed — Physician Decision | 4 | 5
Not completed — Withdrawal by Subject | 1 | 1
Not completed — ineligible | 2 | 2

BASELINE CHARACTERISTICS:
Population: Patients were evaluable for inclusion in the analysis of response if eligible, had an event (relapse, PD, death or secondary malignancy) any time after enrollment, or completed at least 2 courses of Irinotecan/Temozolomide therapy. Patients off therapy before completion of 2 courses by choice or toxicity were not evaluable for response analysis.
Groups:
- Disease Eval by Bone Marrow or MIBG (Irinotecan/Temozolomide): Evaluation by bone marrow or MIBG scan (metaiodobenzylguanidine scan, a radiopharmaceutical). Patients receive irinotecan hydrochloride (10 mg/m2/dose) over 1 hour on days 1-5 and 8-12 and oral temozolomide (100 mg/m2/dose) on days 1-5. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  irinotecan hydrochloride : Given IV
  temozolomide : Given IV
- Total: Total of all reporting groups
Arm/Group | Disease Eval by Bone Marrow or MIBG (Irinotecan/Temozolomide) | Disease Measurable by CT or MRI Scan (Irinotecan/Temozolomide) | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 28 | 30 | 58
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: days] | 1922 [1682 to 2827] | 1562 [1158 to 2648.5] | 1742 [1420 to 2737.75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 26
  Male | 14 | 19 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 4
  Not Hispanic or Latino | 26 | 22 | 48
  Unknown or Not Reported | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 2 | 6
  White | 20 | 21 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 26 | 28 | 54
  Canada | 2 | 2 | 4
  Australia | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response - Complete Response (CR), Very Good Partial Response (VGPR) and Partial Response (PR)
Description: The patient's best overall response obtained during Reporting Periods 1 and 2 will be scored as "best response". Patients enrolled on Stratum 1 with bone marrow disease, a responder has no tumor cells detectable by routine morphology on 2 subsequent bilateral bone marrow aspirates and biopsies done at least 3 weeks apart. For patients enrolled on stratum 1 with MIBG only disease, response will be assessed using the Curie scale. Patients who have complete resolution of all MIBG positive lesions (CR) or resolution of at least one MIBG positive lesion with persistence of other lesions (PR) will be considered responders. For Stratum 2 a responder is defined to be a patient who achieves a best overall response of CR, VGPR or PR from CT/MRI scans from central review using (RECIST) Response Evaluation Criteria in Solid Tumor. A responder is defined to be a patient who achieves a best overall response of CR (Complete Response), VGPR (Very Good Partial Response) or PR (Partial Response).
Time Frame: up to 6 courses of therapy, or about 6 months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Disease Eval by Bone Marrow or MIBG (Irinotecan/Temozolomide) | Disease Measurable by CT or MRI Scan (Irinotecan/Temozolomide)
Number analyzed (Participants) | 27 | 28
participants | 5 | 3

ADVERSE EVENTS:
Time Frame: Duration of protocol therapy, which could be up to about 1 year
Description: Only eligible patients that received at least one dose of protocol therapy are included for Adverse event reporting (there were 2 ineligible patients on Stratum 1 (27 at risk) and 2 ineligible patients on Stratum 2 (28 at risk).
Arm/Group | Disease Eval by Bone Marrow or MIBG (Irinotecan/Temozolomide) | Disease Measurable by CT or MRI Scan (Irinotecan/Temozolomide)
Serious Adverse Events (participants affected / at risk) | 0/27 | 1/28
Other Adverse Events (participants affected / at risk) | 13/27 | 8/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Disease Eval by Bone Marrow or MIBG (Irinotecan/Temozolomide) (N=27) | Disease Measurable by CT or MRI Scan (Irinotecan/Temozolomide) (N=28)
Death not associated with CTCAE term - Disease progression NOS (General disorders) | 0 (0) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Disease Eval by Bone Marrow or MIBG (Irinotecan/Temozolomide) (N=27) | Disease Measurable by CT or MRI Scan (Irinotecan/Temozolomide) (N=28)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 3 | 3
AST: AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 4 | 2
Alkaline phosphatase (Investigations) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 | 0
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 3 | 3
Hemoglobin (Blood and lymphatic system disorders) | 7 | 7
Hyperglycemia: Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 6 | 2
Hypokalemia: Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 4 | 2
Hyponatremia: Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 3 | 4
Leukocytes (total WBC) (Investigations) | 10 | 7
Lymphopenia (Investigations) | 4 | 3
Nausea (Gastrointestinal disorders) | 0 | 3
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 13 | 8
Pain - Abdomen NOS (Gastrointestinal disorders) | 2 | 2
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 4 | 2
Pain - Head/headache (Nervous system disorders) | 2 | 0
Platelets (Investigations) | 7 | 3
Vomiting (Gastrointestinal disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.